CLINICAL TRIAL: NCT05895968
Title: A Controlled Clinical Study on the Safety and Effectiveness of Barb Suture in Obese Patients Undergoing Posterior Cervical Surgery
Brief Title: Researching the Useful of Barb Suture in Obese Patients Undergoing Posterior Cervical Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY20232136-F-1
Record Dates: First submitted 2023-05-25; First posted 2023-06-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2024-05

CONDITIONS: Cervical Spinal Stenosis; Posterior Cervical Spine Surgery; Barbed Suture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Preoperative (No Intervention)
- postoperative (2 weeks) (Experimental)
  Interventions: Procedure: posterior cervical surgery
- postoperative (4 weeks) (Experimental)
  Interventions: Procedure: posterior cervical surgery
- postoperative (3 months) (Experimental)
  Interventions: Procedure: posterior cervical surgery

INTERVENTIONS:
Procedure: posterior cervical surgery — The patients were operated by the posterior cervical surgery, which were used with the barbed to suture the deep fascia.
  Arms: postoperative (2 weeks); postoperative (3 months); postoperative (4 weeks)

SUMMARY:
Through a single-center, exploratory clinical study, the safety and effectiveness of using barb wire in the incision and suture of posterior cervical surgery in obese patients were evaluated, providing a basis for its wide clinical application in posterior cervical surgery.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms and signs of the patients were typical. MRI showed single or multiple central herniation of C3-C7 intervertebral discs or spinal stenosis at corresponding levels, which confirmed cervical myeloid cervical spondylosis or cervical spinal stenosis.
* Preoperative routine tests and examinations showed no contraindications.
* BMI≥28
* Informed consent was obtained from the patient and his family, informed consent was signed, and a complete follow-up was completed after surgery.

Exclusion Criteria:

* A history of wasting diseases associated with malignancy and chemoradiotherapy that may interfere with wound healing
* History of dermatosis
* History of immune system diseases
* History of blood diseases
* Skin injury or defect at the back of the neck
* Severe hypersensitivity
* Cold, fever, trauma or other infections in the week before surgery
* Infectious disease
* Psychosis could not cooperate with follow-up

Ages: 28 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
JOA score change | 3 months after surgery
  JOA score is used to assess the function of spinal cord which is in the form of questionnaires. Postoperative improvement rate = ((postoperative score - preoperative score)/ (17- preoperative score)) X100%. Improvement rate can also correspond to the commonly used efficacy criteria: cure when the improvement rate is 100%, effective when the improvement rate is greater than 60%, effective when 25-60%, and ineffective when less than 25%.
NDI score change | 3 months after surgery
  NDI score is used to assess the disorder of spinal cord which is in the form of questionnaires. Postoperative improvement rate = (total score)/ (numbers of programme X5) X100%. Improvement rate can also correspond to the commonly used efficacy criteria: the improvement rate when 60%-80% means extremely severe dysfunction, when 40%-60% means severe dysfunction, when 20-40% means moderate dysfunction, and when less than 20% means mild dysfunction.
VAS score change | 3 months after surgery
  A Visual Analogue Scale (VAS) is used to measure the amount of pain that a patient feels ranges across a continuum from none to an extreme amount of pain. Using a ruler, the score is determined by measuring the distance (mm) on the 10cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity.

SECONDARY OUTCOMES:
wound infection | 2 weeks after surgery, 4 weeks after surgery, 3 months after surgery
  The presence of wound infection was confirmed through the assessment of the patient's white blood cell count, erythrocyte sedimentation rate, C-reactive protein levels and other relevant biochemical markers. Additionally, signs such as erythema, edema, warmth, tenderness and other related symptoms should be evaluated to determine the presence of wound infection.
wound dehiscence | 2 weeks after surgery, 4 weeks after surgery, 3 months after surgery
  The assessment of wound dehiscence primarily relied on the identification of suture rupture within the wound site through direct visualization.

CONTACTS AND LOCATIONS:
Locations (1):
- Jia Yanyan, Xi'an, Shannxi Province, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chan VWK, Chan PK, Chiu KY, Yan CH, Ng FY. Does Barbed Suture Lower Cost and Improve Outcome in Total Knee Arthroplasty? A Randomized Controlled Trial. J Arthroplasty. 2017 May;32(5):1474-1477. doi: 10.1016/j.arth.2016.12.015. Epub 2016 Dec 21. PMID 28089469
- [Background] Lee SW, Kawai M, Tashiro K, Nomura E, Tokuhara T, Kawashima S, Tanaka R, Uchiyama K. Laparoscopic gastrointestinal anastomoses using knotless barbed absorbable sutures are safe and reproducible: a single-center experience with 242 patients. Jpn J Clin Oncol. 2016 Apr;46(4):329-35. doi: 10.1093/jjco/hyv212. Epub 2016 Jan 26. PMID 26819279
- [Background] Greenberg JA, Einarsson JI. The use of bidirectional barbed suture in laparoscopic myomectomy and total laparoscopic hysterectomy. J Minim Invasive Gynecol. 2008 Sep-Oct;15(5):621-3. doi: 10.1016/j.jmig.2008.06.004. Epub 2008 Jul 10. PMID 18619922
- [Background] Sarsam OM, Dunning J, Pochulu B, Baste JM. Robot-assisted bronchoplasty using continuous barbed sutures. J Vis Surg. 2018 Jan 4;4:3. doi: 10.21037/jovs.2017.12.14. eCollection 2018. PMID 29445589
- [Background] Yang S, Qi-Heng T, Yi-Xin Z. Comparison of Standard Suture vs Barbed Suture for Closing the Porcine Knee Joint: Evaluation of Biomechanical Integrity and Permeability. J Arthroplasty. 2018 Mar;33(3):903-907. doi: 10.1016/j.arth.2017.10.008. Epub 2017 Oct 10. PMID 29103781